CLINICAL TRIAL: NCT02550015
Title: The Effect of High Intensity Interval Training on Maximal Oxygen Uptake and Risk Factors for Recurrent Stroke
Brief Title: High Intensity Interval Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/563
Record Dates: First submitted 2015-09-08; First posted 2015-09-15 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: Exercise training; Oxygen consumption
MeSH Terms: conditions — Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Supervised high intensity interval training (uphill treadmill walking 4 x 4 min at 90-95% of peak heart rate) 3 times weekly for 8 weeks
  Interventions: Behavioral: High intensity interval training
- standard care (Other): Standard clinical follow-up care, including general information about importance of physical activity as part of a healthy lifestyle
  Interventions: Behavioral: General information

INTERVENTIONS:
Behavioral: High intensity interval training — Uphill treadmill walking
  Arms: Training
Behavioral: General information — Standard care
  Arms: standard care

SUMMARY:
The purpose of this study is to examine if high intensity interval training after stroke is more effective than standard care to increase maximal oxygen uptake, reduce known risk factors for recurrent stroke and improve function.

DETAILED DESCRIPTION:
Stroke is a leading cause of adult disability. Well designed studies have shown that the majority of the stroke population have low aerobic capacity and many are inactive. This is negative for their health and well-being. Physical inactivity may increase their risk of having recurrent stroke.

The optimal training mode and intensity to improve aerobic capacity after stroke are not clear. High intensity interval training (ie. 90-95% of peak heart rate) has been proven to be more beneficial than moderate and low intensity exercise in order to improve maximal oxygen uptake in patients with cardiac disease. The response from this training on aerobic capacity and physical function in the stroke population are not known.

ELIGIBILITY:
Inclusion Criteria:

* Approved informed consent
* Independent walking > 2 minutes
* First episode of stroke (ischemic or hemorrhagic)
* Minimum 3 months post-stroke
* Living in the community and able to travel to assessment and training site
* Approval to participate from the study's responsible medical doctor
* Modified Rankin Scale 0-3

Exclusion Criteria:

* Impaired cognitive function to give valid informed consent to participate
* Instability of cardiac conditions (ie. serious rhythm disorder, valve malfunction)
* Other conditions where test of maximal oxygen uptake is contraindicated
* Poorly controlled hypertension (>180/100), measured at rest
* > 5 years post stroke
* Subarachnoid hemorrhage
* Participating in other ongoing intervention study
* Other serious illness influencing testing of cardiorespiratory fitness and function at 1 year follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake | 1 year after inclusion
  A graded treadmill test of maximal oxygen uptake using a breath by breath ergospirometer

SECONDARY OUTCOMES:
Change in blood pressure (systolic and diastolic) | 8 weeks and 12 months after inclusion
  Blood pressure will be measured at rest
Walking speed | 8 weeks and 12 months after inclusion
  Walking speed (in minutes:seconds) will be measured with the 10 meter walk test and the Timed Up and Go test.
Leisure time activity and inactive time | 8 weeks and 12 months after inclusion
  Using the ActivePal monitor attached to the participants non-affected leg information on position, walking and inactive time will be measured during 3 whole consecutive days.
Balance tested with the Bergs Balance Test | 8 weeks and 12 months after inclusion
Change in Blood tests | 8 weeks and 12 months after inclusion
  The following blood tests will be taken: Hemoglobin, HDL, LDL, Cholesterol, Total Cholesterol, C peptides, Triglycerides and HbA1c
Independence assessed by Functional Independence Measure (FIM) | 8 weeks and 12 months after inclusion
Self reported physical activity level assessed by International Physical Activity Questionnaire | 8 weeks and 12 months after inclusion
Cognitive function assessed by Montreal Cognitive Assessment and Trail Making A and B | 8 weeks and 12 months after inclusion
Walking distance | 8 weeks and 12 months after inclusion
  Walking distance (in meters) will be measured with the 6 minute walk test.

OTHER OUTCOMES:
New cardiovascular or cerebrovascular incidents | 8 weeks and 12 months after inclusion
  Gathered from the participants and their electronic journal system
Severity of stroke | 8 weeks and 12 months after inclusion
  The Stroke Impact Scale will be used to evaluate how the stroke has affected the participants' health and life in addition to the National Institute of Health Stroke scale
Anxiety and depression after stroke | 8 weeks and 12 months after inclusion
  Hospital and Anxiety and Depression Scale will be used to get information about the participants level of anxiety and depression
Degree of disability and dependence | 8 weeks and 12 months after inclusion
  Modified Rankin Scale (mRS)
Health status assessed by The Norwegian version of EQ-5D-5L questionnaire | 8 weeks and 12 months after inclusion
Submaximal oxygen consumption during treadmill walking | 8 weeks and 12 months after inclusion
  Oxygen consumption will be measured at a standardized speed and inclination.

CONTACTS AND LOCATIONS:
Overall Officials: Torunn Askim, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Trondheim, Norway

REFERENCES:
- [Result] Gjellesvik TI, Becker F, Tjonna AE, Indredavik B, Nilsen H, Brurok B, Torhaug T, Busuladzic M, Lydersen S, Askim T. Effects of High-Intensity Interval Training After Stroke (the HIIT-Stroke Study): A Multicenter Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Jun;101(6):939-947. doi: 10.1016/j.apmr.2020.02.006. Epub 2020 Mar 4. PMID 32145280